CLINICAL TRIAL: NCT04976309
Title: Interventional, Randomized, Double-blind, Parallel-group, Placebo-controlled Study Investigating the Effect of Lu AG09222 on PACAP38- and VIP-induced Vasodilation, Heart Rate Increase, and Headache in Healthy Subjects
Brief Title: A Single Dose Study of Lu AG09222 in a Headache Model With Healthy Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: H. Lundbeck A/S (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 19734A
Record Dates: First submitted 2021-07-19; First posted 2021-07-26 (Actual); Last update posted 2022-01-19 (Actual); Status verified 2022-01

CONDITIONS: Healthy

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Placebo + saline (Experimental): Placebo, 0.9% normal saline, single dose intravenous infusion over 30 minutes
  Interventions: Drug: Placebo
- Placebo + VIP and PACAP (Experimental): Placebo, 0.9% normal saline, single dose intravenous infusion over 30 minutes
  Interventions: Drug: Placebo
- Lu AG09222 + VIP and PACAP (Experimental): Lu AG09222, single dose intravenous infusion over 30 minutes
  Interventions: Drug: Lu AG09222

INTERVENTIONS:
Drug: Lu AG09222 — Single dose
  Arms: Lu AG09222 + VIP and PACAP
Drug: Placebo — Single dose
  Arms: Placebo + VIP and PACAP; Placebo + saline

SUMMARY:
The purpose of this study is to evaluate how well Lu AG09222 can prevent blood vessel dilation in a headache model.

DETAILED DESCRIPTION:
This study will investigate the effect of preventive treatment with Lu AG09222 on vasodilation, heart rate increase, and headache induced by PACAP and VIP.

Subjects will be randomised to three arms, placebo + saline, placebo + VIP and PACAP, and Lu AG09222 + VIP and PACAP. Subjects who complete the study will attend a safety follow-up visit at 10 to 12 weeks after administration of investigational medicinal product.

ELIGIBILITY:
Inclusion Criteria:

* The subject has a body mass index (BMI) ≥ 18.0 and ≤ 30.0 kg/m2, and a body weight ≥ 45 and ≤ 95 kg at the screening visit.
* The subject is, in the opinion of the investigator, generally healthy based on medical history, a physical examination, vital signs, an ECG, and the results of the clinical chemistry, haematology, urinalysis, serology, and other laboratory tests at screening.

Exclusion Criteria:

* The subject fulfils the diagnostic criteria for a primary headache disorder, or has a first degree relative with a primary headache disorder, according to the International Headache Society (IHS) International Classification of Headache Disorders 3rd edition (ICHD-3), except tension-type headache.
* The subject has or has had tension-type headache more than once per month on average during the 6 months prior to the screening visit.

Other inclusion and exclusion criteria may apply.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 25 (Actual)
Dates: Start 2021-07-15 (Actual); Primary Completion 2021-09-19 (Actual); Study Completion 2021-12-10 (Actual)

PRIMARY OUTCOMES:
Area under the curve (AUC) of change from start of infusion in superficial temporal artery (STA) diameter from 0 to 120 min after start of infusion of PACAP38 | 0 to 120 min after infusion

SECONDARY OUTCOMES:
Change from start of infusion in STA diameter to 60 min after start of infusion of PACAP38 | 0 to 60 min after infusion
Maximum change from start of infusion in STA diameter between 0 and 120 min after start of infusion of PACAP38 | 0 and 120 min after infusion
AUC in change from start of infusion in facial blood flow from 0 to 120 min after start of infusion of PACAP38 | 0 to 120 min after infusion
AUC in change from start of infusion in heart rate from 0 to 120 min after start of infusion of PACAP38 | 0 to 120 min after infusion

CONTACTS AND LOCATIONS:
Overall Officials: Email contact via H. Lundbeck A/S, Study Director — LundbeckClinicalTrials@lundbeck.com
Locations (1):
- Danish Headache Center Rigshospitalet Glostrup, Glostrup Municipality, Denmark

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Rasmussen NB, Deligianni C, Christensen CE, Karlsson WK, Al-Khazali HM, Van de Casteele T, Granhall C, Amin FM, Ashina M. The effect of Lu AG09222 on PACAP38- and VIP-induced vasodilation, heart rate increase, and headache in healthy subjects: an interventional, randomized, double-blind, parallel-group, placebo-controlled study. J Headache Pain. 2023 May 25;24(1):60. doi: 10.1186/s10194-023-01599-w. PMID 37231350